CLINICAL TRIAL: NCT05540197
Title: Arginine-stimulated Indication of Early Outcome After Islet Transplantation
Acronym: ALADDIN
Status: Enrolling by invitation | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Eelco JP de Koning, Prof. Eelco de Koning, Leiden University Medical Center
Other Study IDs: NL79536.058.22
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Islets of Langerhans Transplantation; Diabetes Mellitus; Chronic Pancreatitis
Keywords: total pancreatectomy; autologous islet transplantation; TPIAT; beta-cell function; c-peptide; arginine; mixed meal tolerance test; allogeneic islet transplantation; islet function; ibmir
MeSH Terms: conditions — Diabetes Mellitus; Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma to analyse circulating free DNA, microRNA, T-cell phenotype. Blood cell composition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autologous islet transplantation: Arginine stimulation test: 5 grams of arginine hydrochloride intravenously. Performed at baseline after mixed meal tolerance test (MMTT), performed separately at day -1 or 0, day 1, day 3, day 7 and 3 months, and also at 3 months after MMTT.
- Allogeneic islet transplantation: Arginine stimulation test: 5 grams of arginine hydrochloride intravenously. Performed at day -1 or 0, day 1, day 3, day 7, 3 months and at 3 months after MMTT.

SUMMARY:
Through islet transplantation, functional β-cell mass can be restored. Allogeneic islet transplantation is a treatment modality for a select group of patients with complicated type 1 diabetes mellitus. For patients undergoing (partial) pancreas resection, autologous islet transplantation may help prevent complicated diabetes. Up until now, no studies have been performed on early islet graft function in the first week after transplantation. Early graft function may be a predictor for estimating long-term islet graft success.

Arginine can excite β-cells to release insulin. It can thus provide an estimate of β-cell secretory capacity and can be used as an alternative to (oral) glucose tolerance tests. In this study, we aim to find a predictor model for islet graft function by assessing peak C-peptide after arginine stimulus in the early post-transplantation phase.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or older
* Currently on the LUMC waiting list for allogeneic or autologous islet transplantation
* Willing to use a flash glucose monitoring (FGM) system in the two weeks prior to transplantation

Exclusion Criteria:

* Patients who are pregnant
* Patients with known hypersensitivity to arginine

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving allogeneic or autologous islet transplants.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Early islet graft function | Day 3
  Peak C-peptide during AST at day 3
Early islet graft function | Month 3
  AUC C-peptide during MMTT at 3 months

SECONDARY OUTCOMES:
Early islet graft function | Up to 3 months
  Peak C-peptide during AST and MMTT (other than primary)
Early islet graft function | Up to 3 months
  AUC C-peptide during AST and MMTT (other than primary)
Insulin secretory capacity | Up to 3 months
  Relationship between in vitro secretion and in vivo secretion
Beta-cell death | Up to 3 months
  Circulating free INS DNA (INS cfDNA)
Beta-cell death | Up to 3 months
  insulin - proinsulin ratio
Beta-cell death | Up to 3 months
  Plasma circulating microRNA
Complement factors | Up to 3 months
  Markers of complement activation
Immunological markers | Up to 3 months
  Peripheral blood mononuclear cell (PBMC) composition
Immunological markers | Up to 3 months
  T-cell phenotyping
Beta cell graft function | Up to 3 months
  Time in range, time below range, time above range as measured by Flash Glucose Monitoring (FGM) or Continuous Glucose Monitoring (CGM)
Beta cell graft function | 3 months
  assessed by Igls 2.0 criteria
Treatment success | 3 months
  assessed by Igls 2.0 criteria
Beta cell graft function | Up to 3 months
  Amount of severe hypoglycaemic events
Beta cell graft function | Up to 3 months
  Insulin requirements (IU/kg/day)
Glycemic control | Up to 3 months
  HbA1c (mmol/mol)
Coagulation markers | Up to 3 months
  Markers indicative for activation of the coagulation cascade
Insulin concentration | Before the islet transplantation
  Concentration of insulin in the islet product

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Eelco de Koning, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided